CLINICAL TRIAL: NCT01587183
Title: Running Against Prehypertension Trial (RAPT): A Pilot Randomized Controlled Trial
Brief Title: Running Against Prehypertension Trial (RAPT): A Pilot Trial
Acronym: RAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12-08425
Record Dates: First submitted 2012-03-29; First posted 2012-04-30 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Prehypertension
Keywords: Running; Blood pressure
MeSH Terms: conditions — Prehypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Educational materials control (Other): Enhanced usual care
  Interventions: Behavioral: Educational material control
- Group running style B (Active Comparator): Basic running instruction using group based training.
  Interventions: Behavioral: Group running style B
- Group running style A (Experimental): Form focused running instruction using group based training.
  Interventions: Behavioral: Group running style A

INTERVENTIONS:
Behavioral: Educational material control — Participants will be given educational materials on starting a running program using a run/walk approach.
  Arms: Educational materials control
Behavioral: Group running style B — Participants will attend a 4 hour group based training and 3, 2 hour follow up trainings.
  Arms: Group running style B
Behavioral: Group running style A — Participants will attend a 4 hour group based training and 3, 2 hour follow up trainings.
  Arms: Group running style A

SUMMARY:
This study will test strategies to help people with prehypertension adopt a running program to reduce their blood pressure in the long term. This study will be a 12 week intervention of about 40 participants randomized to running educational material, group based running instruction, or group based running instruction focused on form and all given the option to use the supplemental mHealth intervention. The purpose of this study is to collect feasibility, acceptability and preliminary efficacy data in preparation for a larger planned NIH-R01 study.

DETAILED DESCRIPTION:
The UCSF Osher Center for Integrative Medicine has increasingly been investigating lifestyle interventions and their upstream approach to improving health and well-being. Many such lifestyle interventions address health risk nonpharmacologically and present participants with the opportunity to change their overall trajectory of health. Exercise interventions are of particular interest based on evidence of numerous physical and mental health benefits. Our target population in the Running Against Prehypertension Trial (RAPT) was people with upper range prehypertension. By adopting and maintaining a running program, these individuals who are at a high risk of hypertension can avoid a lifetime of medication and chronic disease. The objective of RAPT was to collect feasibility, acceptability and preliminary efficacy data over a 12 week period on a running program aimed at teaching a natural running form called ChiRunning that used the mindful movement principles of Tai Chi. By using this natural running form, participants may increase satisfaction and decrease rates of injury towards greater adherence to the program. Participants were randomized to one of three study arms: 1) intervention, 8 weeks of group training in form focused ChiRunning; 2) active control, 8 weeks of group training focused on conventional running excluding form; or 3) usual care, a self-directed training with educational materials.

ELIGIBILITY:
Inclusion Criteria:

* The target population for our proposed study is adults with upper range prehypertension defined by systolic blood pressure in the range of 130-144mmHg or diastolic blood pressure range in the range of 85-94mmHg.
* Potential participants will have two to three blood pressure screening measurements at least one day apart taken to screen for eligibility.
* Participants also must not be currently taking antihypertensive medications and must live in the San Francisco Bay Area.

Exclusion Criteria:

1. Inability to provide informed consent
2. Age < 18 years
3. Inability to run continuously for 5 minutes (required for the gait analysis)
4. A substance or alcohol abuse, mental health, or medical condition that, in the opinion of investigators, will make it difficult for the potential subject to participate in the group intervention
5. A history of cardiovascular disease or coronary artery disease including acute coronary syndrome, heart failure, severe aortic stenosis, acute infection or fever, or resting tachycardia (> 100 bpm)
6. A history of cardiac procedures including coronary artery bypass graft, angioplasty or stent placement.
7. Typical or atypical angina
8. Arrhythmia, alcoholism or other condition that makes accurate BP measurement difficult
9. A diagnosis of diabetes, chronic kidney disease or other condition indicating medication for SBP < 140mmHg
10. Non-English speaking (group training will be given in English)
11. Pregnant or planning to get pregnant during the study period
12. Unwillingness or inability to commit to run/walking up to 30 minutes three times per week
13. Plans to move from the San Francisco Bay area during the study time period
14. Currently exercising at vigorous intensity for greater than 90 minutes per week. Vigorous intensity exercise may include race walking, jogging, running, hiking, swimming laps, or bicycling ≥ 10 miles per hour.
15. BMI > 30

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment and retention | At the end of the 8 week recruitment period
  We will determine feasibility associated with recruitment n by recruiting and retaining at least 75% of our intended sample.
Feasibility and acceptability of study protocol and materials | At the end of the 12 week study
  We will conduct both qualitative and quantitative analysis of the evaluations provided by participants to improve study protocol and materials and to indicate feasibility and acceptability of the study content. We will consider at least 75% of participants being "satisfied" or higher in the overall study evaluation to indicate acceptability of the study materials. We will consider completing at least 75% of the intended gait analyses and feedback from the lab specialists to indicate feasibility and a "satisfied" or higher score by at least 75% of participants as being acceptable.
Preliminary efficacy data on changes in blood pressure | Change in systolic and diastolic blood pressure from baseline at the end of the 12 week study
  For the preliminary efficacy data we will compare systolic and diastolic blood pressure changes between baseline and post intervention to determine effect size to make sample size calculations for a larger planned trial.

SECONDARY OUTCOMES:
Preliminary efficacy data on injury incidence | At the end of the 12 week study
  For the preliminary efficacy data on injury incidence across the three study groups. Data on injury incidence will be collected using the training diary questions about whether a run was missed due to injury.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly McDermott, PhD, Principal Investigator — University of California, San Francisco; Fredrick Hecht, MD MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Osher Center for Integrative Medicine, San Francisco, California, United States

REFERENCES:
- [Derived] McDermott K, Kumar D, Goldman V, Feng H, Mehling W, Moskowitz JT, Souza RB, Hecht FM. Training in ChiRunning to reduce blood pressure: a randomized controlled pilot study. BMC Complement Altern Med. 2015 Oct 15;15:368. doi: 10.1186/s12906-015-0895-x. PMID 26471194
- [Derived] Kumar D, McDermott K, Feng H, Goldman V, Luke A, Souza RB, Hecht FM. Effects of Form-Focused Training on Running Biomechanics: A Pilot Randomized Trial in Untrained Individuals. PM R. 2015 Aug;7(8):814-822. doi: 10.1016/j.pmrj.2015.01.010. Epub 2015 Jan 26. PMID 25633634